CLINICAL TRIAL: NCT06196801
Title: Efficacy of Triple-Combination Therapy in Severe Pulmonary Arterial Hypertension Associated Congenital Heart Diseases
Brief Title: Efficacy of Triple-Combination Therapy in Severe PAH-CHD
Status: Active, not recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Caojin, MD, Chief Physician, Guangdong Provincial People's Hospital
Other Study IDs: Triple CHD PAH 2021
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Triple Combination therapy
  Interventions: Drug: Triple-combination therapy

INTERVENTIONS:
Drug: Triple-combination therapy — phosphodiesterase 5 inhibitors, endothelin receptor antagonist, and parenteral prostacyclin

SUMMARY:
Congenital heart disease (CHD) is a leading cause of pulmonary arterial hypertension (PAH) worldwide. Treatment for PAH associated with CHD (PAH-CHD) depends on the defect's type, size, and hemodynamic impact. For those with CHD correction indications, early defect repair or interventional closure is crucial to prevent irreversible pulmonary vascular remodeling due to prolonged exposure to a left-to-right shunt.

Current guidelines recommend triple-combination therapy, including phosphodiesterase 5 inhibitors, endothelin receptor antagonist, and parenteral prostacyclin, for patients with intermediate-high or high risk. Recent studies suggest that patients with PAH-CHD and borderline hemodynamics might regain eligibility for surgery after targeted vasodilatory treatment. Consequently, early initiation of triple-combination therapy may be critical for severe PAH-CHD patients to restore their surgical or interventional closure eligibility. Therefore, we conducted this prospective study to assess the effectiveness of triple-combination therapy in severe PAH-CHD cases.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with congenital heart diseases (CHD) and associated pulmonary arterial hypertension (PAH)
2. Subject is under borderline hemodynamics status and ineligible for congenital heart diseases closure, confirmed by RHC: Qp/Qs：< 1.5, Rp/Rs > 0.3 and PVR > 5 Wood units
3. Subject signs an informed Consent Form and is willing to participate in follow-up visits

Exclusion Criteria:

1. Subject is diagnosed with other etiology of pulmonary arterial hypertension, e.g. left heart diseases associated pulmonary arterial hypertension.
2. Subject is diagnosed with other types of PAH-CHD, e.g. Eisenmenger syndrome, PAH with small/coincidentalb defects
3. Subject had cerebral hemorrhage, bleeding events in other organs within 3 months or was in high risk of bleeding.
4. Subject is diagnosed of hepatic insufficiency: ALT or AST>3×ULN at the screening visit.
5. Subject is diagnosed of moderate to severe renal insufficiency: eGFR<30ml/min/1.73m2 at the screening visit.
6. Subject has uncontrolled arrhythmia with clinical significance within 90 days.
7. Subject is diagnosed of the following diseases or received following medical interventions with 90 days: unstable angina, severe coronary atherosclerosis or myocardial infarction, cerebrovascular disease, deep vein thrombosis, pulmonary embolism, percutaneous coronary intervention, coronary artery bypass grafting, carotid artery intervention, peripheral artery intervention.
8. Subject is diagnosed of malignant tumor (exception: tumors that have been cured and have not recurred in the last 5 years, basal cell and squamous cell skin cancers that have been completely resected, and cancers of any type in situ that have been completely resected)
9. Subject cannot follow the study procedure due to other acute or chronic diseases.
10. Subject is under other RCT.
11. Subject has a life expectancy <1 year.
12. Subject cannot follow the study procedure due to other reasons in the opinion of the investigators. (alcoholic, drug abuse, lack of compliance)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patints diagnosed of congenital heart diseases with severe pulmonary arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary hemodynamics | 6 months,12 months
  comparison of hemodynamics at baseline, before and after surgery/intervention, assessed by RHC

SECONDARY OUTCOMES:
Pulmonary hemodynamics | perioperative period
Vasodilators average usage and compliance | 6 months, 12 months
Surgery success rate and adverse event | surgery perioperative period
Other monitoring data | surgery perioperative period
Other examination results | surgery perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Cardiovascular Institute, Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No